CLINICAL TRIAL: NCT04677946
Title: Dietary Oil to Improve Sleep Quality: SNACk Study
Brief Title: Dietary Oil to Improve Sleep Quality
Acronym: SNACk
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Martha Belury, Associate Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019H0327
Record Dates: First submitted 2020-09-18; First posted 2020-12-21 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Insomnia Type; Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Cookie Group (Experimental): All participants in the study
  Interventions: Other: High Linoleic Acid Healthy Cookies

INTERVENTIONS:
Other: High Linoleic Acid Healthy Cookies — High Linoleic Acid Healthy Cookies (containing about 9g of linoleic acid) 1 per day for 8 weeks

SUMMARY:
The purpose of this study is to identify if healthy cookies high in linoleic acid can change sleep quality and sleep architecture, blood fatty acid composition and be consumed with high compliance after eight weeks of consumption. The hypothesis is that consumption of healthy cookies for 8 weeks will improve sleep quality, increase linoleic acid in the blood and be consumed with greater than 80% compliance.

DETAILED DESCRIPTION:
Overall, linoleic acid has many health benefits including altering body composition and energy metabolism, but is not clear if linoleic acid consumption can influence sleep quality.

The investigators plan to test the central hypothesis and accomplish the overall objective of this research by pursuing the following specific aims

Aim 1) To determine the effect of healthy cookies made with linoleic acid-rich oil on measures of sleep quality and sleep architecture in overweight adults

Aim 2) To determine the effect on plasma fatty acid composition and markers of circadian rhythm in peripheral blood mononuclear cells (PBMC) after four and eight weeks of consuming one healthy cookie per day

Aim 3) To measure the effect of healthy cookies made with LA-oil on change of lipidomic profiles of plasma and PBMC after four and eight weeks of consumption

Aim 4) To determine the feasibility of adherence to consuming 1 healthy cookie per day in place of snack for eight weeks

ELIGIBILITY:
Inclusion Criteria:

* Overweight (BMI ≥25 and <38)
* Nonsmoker
* Insomnia severity index score ≥8

Exclusion Criteria:

* Current or previous diagnosis of diabetes, heart (including stroke or heart attack), kidney, liver or circulatory diseases and/or current treatment for cancer
* Gastrointestinal diseases or disorders (including pancreatic) or gastric bypass surgery
* Food Allergy or Intolerance
* Any dietary restriction where consumption of these healthy cookies or any ingredient would be contraindicated
* Use of medications where consuming the healthy cookies would be contraindicated
* Usage of sleep aid (prescription medication(s)) for insomnia
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2027-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Changes in sleep quality using the Pittsburgh Sleep quality index, PROMIS Sleep questionnaire, and insomnia severity index questionnaire | Week 0, week 4 and week 8
  Changes in global sleep quality scores using the Pittsburgh sleep quality index PROMIS Sleep questionnaire, and insomnia severity index measurements
Feasibility of daily healthy cookie consumption | Week 8
  Percent of healthy cookies consumed
Changes in blood fatty acids | Week 0, week 4 and week 8
  Changes in linoleic acid levels in the blood
Changes in markers of circadian rhythm | Week 0, week 4 and week 8
  Changes in mRNA expression of genes related to circadian rhythm in peripheral blood mononuclear cells
Changes in blood lipidomic profiles | Week 0, week 4 and week 8
  Changes in linoleic acid oxylipins in plasma and cardiolipin in peripheral blood mononuclear cells
Changes in activity during waking and sleeping hours using an actigraph | Week 0, week 4 and week 8
  Changes in activity during waking and sleeping hours each day will be measured using actigraphy
Changes in sleep electroencephalography (EEG) | Week 0, week 4 and week 8
  Changes in sleep EEG will be measured to determine sleep efficiency, arousal index, total sleep time

SECONDARY OUTCOMES:
Changes in body shape using body mass index (calculated using height and weight) and abdominal thickness | Week 0 and week 8
  Changes in body mass index and sagittal diameter
Changes in marker of glycemia | Week 0, week 4 and week 8
  Changes in glucose and insulin
Changes in markers of muscle function using gait speed and grip strength | Week 0 and week 8
  Changes in grip (hand strength) and gait (walking) speed
Changes in markers of inflammation | Week 0, week 4 and week 8
  Changes in interleukin 6, tumor necrosis factor receptor 2, C-reactive protein